CLINICAL TRIAL: NCT06145685
Title: Effect of Smoking Cessation on Salivary IL-1β and PGE-2 Levels Following Non-Surgical Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Collaborators: Ain Shams University (Other); Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Ahmed Y Gamal, Professor of Oral Medicine, Periodontology and Oral Diagnosis, Faculty of Dentistry, Ain Shams University. Professor of Periodontology, College of Oral and Dental Surgery, Misr University for Science and Technology., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-2014 OMD
Record Dates: First submitted 2023-11-12; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Periodontal Diseases; Smoking Cessation
Keywords: Smoking Cessation; Periodontal Diseases; Inflammatory Markers; Interleukin-1beta; Prostaglandin E2; Non-surgical therapy; Smoking
MeSH Terms: conditions — Periodontal Diseases; Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Previous smokers - Minimally invasive (Active Comparator): Minimally invasive non-surgical periodontal treatment
  Interventions: Procedure: Minimally invasive non-surgical periodontal therapy
- Previous smokers - Conventional (Active Comparator): Conventional non-surgical periodontal treatment
  Interventions: Procedure: Conventional non-surgical periodontal therapy
- Smoker (Active Comparator): Conventional non-surgical periodontal treatment
  Interventions: Procedure: Conventional non-surgical periodontal therapy
- Non-smoker (Active Comparator): Conventional non-surgical periodontal treatment
  Interventions: Procedure: Conventional non-surgical periodontal therapy

INTERVENTIONS:
Procedure: Minimally invasive non-surgical periodontal therapy — Minimally invasive non-surgical periodontal therapy
  Arms: Previous smokers - Minimally invasive
Procedure: Conventional non-surgical periodontal therapy — Conventional non-surgical periodontal therapy
  Arms: Non-smoker; Previous smokers - Conventional; Smoker

SUMMARY:
The aim of this study is to evaluate the effect of smoking cessation on inflammatory markers following non-surgical treatment of periodontal disease. This is to assess the period of smoking abstinence needed before any periodontal surgery in order to reverse the negative effects of the reported increased levels of inflammatory markers (IL-1β and PGE2 in this study) associated with smoking on the healing and the periodontium.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced chronic periodontitis upon clinical examination with clinical attachment loss (CAL) more than 5 mm.
* Patients willing to quit smoking to be included in two groups, while patients unwilling to quit smoking to be included in the third group, and the non-smokers as the fourth group.

Exclusion Criteria:

* Any systemic illness known to affect the outcome.
* Systemic antimicrobial or anti-inflammatory drug therapy within the last 3 months prior to the study.
* Patients unable to perform routine oral hygiene procedures.
* Patients using other forms of tobacco.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Levels of Prostaglandin E2 | Baseline and 2 months
  Salivary biochemical analysis
Interleukin 1 beta (in PG/ml) | Baseline and 2 months
  Salivary biochemical analysis

SECONDARY OUTCOMES:
Pocket depth (in mm) | Baseline and 9 months
  Periodontal clinical parameter
clinical attachment level (in mm) | Baseline and 9 months
  Periodontal clinical parameter
bone gain (in mm) | Baseline and 9 months
  Periodontal clinical parameter
Plaque index (scores) | Baseline and 9 months
  Periodontal clinical parameters
Periodontal clinical parameters | Baseline and 9 months
  Gingival index (scores)

CONTACTS AND LOCATIONS:
Overall Officials: Noura M ElShiaty, Dr., Principal Investigator — Master Degree in Diagnosis, Oral Medicine and Periodontology - Faculty of Dentistry - Ain Shams University, Membership of the Faculty of Dental Surgery of The Royal College of Surgeons of Edinburgh; Fatma H El-Demerdash, Associate Professor, Study Director — Associate Professor of Periodontology, Oral Medicine and Diagnosis - Faculty of Dentistry - Ain Shams University, Associate Professor of Oral Medicine and Periodontology - Faculty of Oral and Dental Medicine - Misr International University; Hussien Elkholy, Associate Professor, Study Director — Associate Professor of Psychiatry - Faculty of Medicine - Ain Shams University; Ahmed Y Gamal, Professor, Study Director — Professor of Oral Medicine, Periodontology and Oral Diagnosis - Faculty of Dentistry - Ain Shams University, Professor of Periodontology - College of Oral and Dental Surgery - Misr University for Science and Technology
Locations (1):
- Ain Shams University, Cairo, Egypt